CLINICAL TRIAL: NCT00908687
Title: A Randomized Blinded, LT Dose-ranging Study to Assess the Immunogenicity and Safety of Different Doses of LT Adjuvant Patch Administered in Conjunction With Different Doses of Inactivated Influenza A/H5N1 Vaccine in Healthy Adults
Brief Title: A/H5N1/LT Dose Ranging Study
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Intercell USA, Inc. (Industry)
Collaborators: Department of Health and Human Services (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: PLA201; HHSO100200700031C
Record Dates: First submitted 2009-05-22; First posted 2009-05-27 (Estimated); Results first posted 2014-03-13 (Estimated); Last update posted 2021-12-10 (Actual); Status verified 2021-12

CONDITIONS: Pandemic Influenza

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (6):
- Group 1: 30 µg HA, no LT patch (Experimental): A/H5N1 Vaccine 30 µg HA i.m. on Day 0
  Interventions: Biological: A/H5N1
- Group 2: 30 µg HA + 50 µg LT patch (Experimental): A/H5N1 Vaccine 30 µg HA i.m. + LT adjuvant patch containing 50 µg of LT on Day 0
  Interventions: Biological: A/H5N1; Biological: LT Adjuvant Patch
- Group 3: 30 µg HA + 100 µg LT patch (Experimental): A/H5N1 Vaccine 30 µg HA i.m. + LT adjuvant patch containing 100 µg of LT on Day 0
  Interventions: Biological: A/H5N1; Biological: LT Adjuvant Patch
- Group 4: 45 µg HA, no LT patch (Experimental): A/H5N1 Vaccine 45 µg HA i.m. on Day 0
  Interventions: Biological: A/H5N1
- Group 5: 45 µg HA + 50 µg LT patch (Experimental): A/H5N1 Vaccine 45 µg HA i.m. + LT adjuvant patch containing 50 µg of LT on Day 0
  Interventions: Biological: A/H5N1; Biological: LT Adjuvant Patch
- Group 6: 45 µg HA + 100 µg LT patch (Experimental): A/H5N1 Vaccine 45 µg HA i.m. + LT adjuvant patch containing 100 µg of LT on Day 0
  Interventions: Biological: A/H5N1; Biological: LT Adjuvant Patch

INTERVENTIONS:
Biological: A/H5N1 — A/H5N1 Low Dose
  Arms: Group 1: 30 µg HA, no LT patch; Group 2: 30 µg HA + 50 µg LT patch; Group 3: 30 µg HA + 100 µg LT patch
Biological: A/H5N1 — A/H5N1 High Dose
  Arms: Group 4: 45 µg HA, no LT patch; Group 5: 45 µg HA + 50 µg LT patch; Group 6: 45 µg HA + 100 µg LT patch
Biological: LT Adjuvant Patch — LT Adjuvant Patch Low Dose
  Arms: Group 2: 30 µg HA + 50 µg LT patch; Group 5: 45 µg HA + 50 µg LT patch
Biological: LT Adjuvant Patch — LT Adjuvant Patch High Dose
  Arms: Group 3: 30 µg HA + 100 µg LT patch; Group 6: 45 µg HA + 100 µg LT patch

SUMMARY:
This is a Phase 2, randomized, blinded, clinical trial. Up to 500 eligible subjects will be enrolled and randomized in a 1:2:2:1:2:2 ratio into one of six groups, and vaccinated in this study. Subjects will receive an intramuscular injection of the influenza A/H5N1 (low or high dose) on Day 0 with or without a patch (low or high dose).

ELIGIBILITY:
Inclusion Criteria:

* Healthy adult male or females 18 to 49 years of age (inclusive)
* Signed Informed Consent
* Women who are not post-menopausal or surgically sterile must have a negative serum or urine pregnancy test at screening and within 24 hours of vaccination with understanding (through informed Consent process) to not become pregnant over the duration of the study, and must agree to employ an effective form of birth control for the duration of the study. Acceptable forms of birth control are: abstinence, hormonal contraceptives (oral, injectable, implant, patch, ring), double-barrier contraceptives (condom or diaphragm, with spermicide) and IUD

Exclusion Criteria:

* Clinically significant laboratory abnormalities at screening
* Abnormalities at physical examination [as determined by the Toxicity Grading Scale (grade 1-4)]
* Known allergies to any component of the vaccine
* Known egg protein allergy
* Known allergies to adhesives
* Known disturbance of coagulation
* Participated in research involving investigational product within 45 days before planned date of vaccination
* Donated or received blood or blood products such as plasma within the past 45 days
* Received any licensed vaccines within 2 weeks (for inactivated vaccines) or 4 weeks (for live vaccines) prior to planned date of vaccination
* Ever received investigational enterotoxigenic E. coli, or LT (R192G) or NasalFlu, Berna Biotech Ltd
* Ever received cholera toxin or vaccine (e.g. Orochol, Dukoral)
* History of abdominal surgery (excluding C-Section, hysterectomy, cosmetic surgery, liposuction, appendectomy, cholecystectomy, ventral hernia repair, and other surgeries not pertaining to gastrointestinal problems) or history of, or recent acute gastrointestinal (GI) illness
* Previous vaccination with a pandemic vaccine or previous proven contact with A/H5N1 wild type virus (contact with an individual with laboratory-confirmed A/H5N1 infection or contact with an animal which died as a result of A/H5N1 infection)
* Recent or regular use of oral, topical or injected steroid medications within 45 days prior to vaccination
* Use of immunosuppressive systemic steroid medications including inhaled steroids within three months prior to vaccination
* Comorbid conditions or treatments that are immunosuppressive, including cancer, diabetes, and end-stage renal disease, as determined by the Investigator
* Positive serology for HIV-1, HIV-2, HBsAg, or HCV
* History of severe atopy
* Medical history of acute or chronic skin disease at vaccination area
* Active skin allergy
* Signs of acute skin infection, sunburn or skin abnormalities at the vaccination area including fungal infections, severe acne, active contact dermatitis, or a history of keloid formation
* Hirsute (significant amount of hair) at vaccination area
* Artificial tanning (UV radiation) over the duration of the study including the screening period
* Visible tattoos or marks (tattoos/scars) at the vaccination area that would prevent appropriate dermatologic monitoring of the vaccination site
* Fever greater than or equal to 38.0°C (100.4°F) at the time of planned vaccination
* Suspicion of or recent history (within one year of planned vaccination) of alcohol or substance abuse
* Women who are pregnant or breastfeeding
* Acute illness at screening or at baseline
* Ever had a serious reaction to prior influenza vaccination
* Developed a neurological disorder (such as Guillian Barré syndrome) in the six weeks following a previous influenza vaccination
* Medical history of achlorhydria
* Employee of the investigational site or sponsor
* History of employment in bird or poultry industries or considerable exposure to birds (e.g. poultry or avian veterinarians, bird breeders, poultry butchers and/or culler, etc.)

Ages: 18 Years to 49 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 500 (Actual)
Dates: Start 2009-05; Primary Completion 2010-01 (Actual); Study Completion 2011-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Eric Sheldon, MD, Principal Investigator — Miami Research Associates
Locations (6):
- United States (6):
  - Advanced Clinical Research Institute, Anaheim, California
  - Solano Clinical Research, Vallejo, California
  - Miami Research Associates, Miami, Florida
  - Accelovance, South Bend, Indiana
  - Johnson County Clinical Trials, Lenexa, Kansas
  - Jean Brown Research, Salt Lake City, Utah

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Group 1: 30 µg HA, no LT Patch | Group 2: 30 µg HA + 50 µg LT Patch | Group 3: 30 µg HA + 100 µg LT Patch | Group 4: 45 µg HA, no LT Patch | Group 5: 45 µg HA + 50 µg LT Patch | Group 6: 45 µg HA + 100 µg LT Patch
Started | 50 | 100 | 102 | 50 | 98 | 100
Completed | 49 | 99 | 99 | 47 | 94 | 94
Not Completed | 1 | 1 | 3 | 3 | 4 | 6

BASELINE CHARACTERISTICS:
Population: safety population: all subjects with signed Informed Consent who have received investigational product
Groups:
- Total: Total of all reporting groups
Arm/Group | Group 1: 30 µg HA, no LT Patch | Group 2: 30 µg HA + 50 µg LT Patch | Group 3: 30 µg HA + 100 µg LT Patch | Group 4: 45 µg HA, no LT Patch | Group 5: 45 µg HA + 50 µg LT Patch | Group 6: 45 µg HA + 100 µg LT Patch | Total
Number analyzed (Participants) | 50 | 100 | 102 | 50 | 98 | 100 | 500
Age, Continuous [Mean (Standard Deviation); unit: years] | 30.9 (9.7) | 29.8 (9.6) | 31.3 (10.4) | 30.5 (8.7) | 28.1 (8.2) | 30.8 (8.3) | 30.1 (9.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 29 | 54 | 61 | 25 | 53 | 64 | 286
  Male | 21 | 46 | 41 | 25 | 45 | 36 | 214

OUTCOME MEASURES:

1. Primary Outcome: Assess the Proportion of Subjects in Each Dose Group Achieving Seroconversion and Seroprotection for HI Antibody Titer Through Day 28.
Description: Seroconversion is defined as either 1) baseline HI titer < 1:10 and a post-vaccination HI titer ≥ 1:40, or 2) baseline HI titer ≥ 1:10 and a minimum four-fold rise. Seroprotection is defined as a post-vaccination HI antibody titer ≥ 1:40. FDA/EMEA criterion for seroconversion was to meet or exceed 40%. FDA/EMEA criterion for seroprotection was to meet or exceed 70%.
Time Frame: Day 28
Population: Primary Immunogenicity Evaluable Population (PIEP): all subjects who were consented, randomized, received the assigned treatment, had HI assay results at all the following time points: baseline (Day 0), Day 21 and Day 28, and did not have any major protocol deviations
Measure: Number (95% Confidence Interval); unit: percentage of subjects
Arm/Group | Group 1: 30 µg HA, no LT Patch | Group 2: 30 µg HA + 50 µg LT Patch | Group 3: 30 µg HA + 100 µg LT Patch | Group 4: 45 µg HA, no LT Patch | Group 5: 45 µg HA + 50 µg LT Patch | Group 6: 45 µg HA + 100 µg LT Patch
Number analyzed (Participants) | 49 | 98 | 101 | 50 | 96 | 94
percentage of subjects
  HI Seroconversion Rates | 35.4 [22.2 to 50.5] | 47.4 [37.2 to 57.8] | 37.6 [28.2 to 47.8] | 53.1 [38.3 to 67.5] | 50.5 [40.1 to 61.0] | 50.0 [39.5 to 60.5]
  HI Seroprotection Rates | 35.4 [22.2 to 50.5] | 47.4 [37.2 to 57.8] | 37.6 [28.2 to 47.8] | 55.1 [40.2 to 69.3] | 53.7 [43.2 to 64.0] | 50.0 [39.5 to 60.5]

2. Secondary Outcome: Safety of A/H5N1 Vaccine IM Injection With and Without an LT Adjuvant Patch
Time Frame: 6 months
Measure: Number; unit: Number of Events
Arm/Group | Group 1: 30 µg HA, no LT Patch | Group 2: 30 µg HA + 50 µg LT Patch | Group 3: 30 µg HA + 100 µg LT Patch | Group 4: 45 µg HA, no LT Patch | Group 5: 45 µg HA + 50 µg LT Patch | Group 6: 45 µg HA + 100 µg LT Patch
Number analyzed (Participants) | 50 | 100 | 102 | 50 | 98 | 100
Number of Events
  All AEs | 70 | 484 | 507 | 136 | 516 | 471
  Local AEs | 19 | 309 | 358 | 37 | 361 | 337
  Systemic AEs | 51 | 175 | 149 | 99 | 155 | 134
  All Severe AEs | 4 | 28 | 13 | 6 | 26 | 28
  Severe Local AEs | 0 | 18 | 11 | 0 | 18 | 21
  Related Severe Local AEs | 0 | 18 | 11 | 0 | 18 | 21
  Severe Systemic AEs | 4 | 10 | 2 | 6 | 8 | 7
  Related Severe Systemic AEs | 2 | 4 | 0 | 1 | 4 | 3
  All Serious AEs | 0 | 0 | 1 | 0 | 1 | 1
  Serious Local AEs | 0 | 0 | 0 | 0 | 0 | 0
  Serious Systemic AEs | 0 | 0 | 1 | 0 | 1 | 1

3. Secondary Outcome: Evaluate Treatment Group HI Responses Against US FDA Guidance for Industry: Clinical Data Needed to Support the Licensure of Pandemic Influenza Vaccines (May 2007) and EMA CPMP/BWP/214/96 Criteria for Immunogenicity
Time Frame: Day 28
Measure: Geometric Mean (95% Confidence Interval); unit: fold increase of Geometric Mean Titers
Arm/Group | Group 1: 30 µg HA, no LT Patch | Group 2: 30 µg HA + 50 µg LT Patch | Group 3: 30 µg HA + 100 µg LT Patch | Group 4: 45 µg HA, no LT Patch | Group 5: 45 µg HA + 50 µg LT Patch | Group 6: 45 µg HA + 100 µg LT Patch
Number analyzed (Participants) | 49 | 98 | 101 | 50 | 96 | 94
fold increase of Geometric Mean Titers | 7.1 [4.8 to 10.5] | 8.4 [6.2 to 11.3] | 8.6 [6.4 to 11.6] | 12.7 [8.5 to 19.2] | 10.7 [8.0 to 14.2] | 13.5 [9.7 to 18.7]

ADVERSE EVENTS:
Arm/Group | Group 1: 30 µg HA, no LT Patch | Group 2: 30 µg HA + 50 µg LT Patch | Group 3: 30 µg HA + 100 µg LT Patch | Group 4: 45 µg HA, no LT Patch | Group 5: 45 µg HA + 50 µg LT Patch | Group 6: 45 µg HA + 100 µg LT Patch
Serious Adverse Events (participants affected / at risk) | 0/50 | 0/100 | 1/102 | 0/50 | 1/98 | 1/100
Other Adverse Events (participants affected / at risk) | 31/50 | 86/100 | 86/102 | 36/50 | 87/98 | 85/100
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Group 1: 30 µg HA, no LT Patch (N=50) | Group 2: 30 µg HA + 50 µg LT Patch (N=100) | Group 3: 30 µg HA + 100 µg LT Patch (N=102) | Group 4: 45 µg HA, no LT Patch (N=50) | Group 5: 45 µg HA + 50 µg LT Patch (N=98) | Group 6: 45 µg HA + 100 µg LT Patch (N=100)
Acute myocardial infarction (Cardiac disorders) | 0 | 0 | 0 | 0 | 1 | 0
Adenomyosis (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 1
Hypotension (Vascular disorders) | 0 | 0 | 1 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Group 1: 30 µg HA, no LT Patch (N=50) | Group 2: 30 µg HA + 50 µg LT Patch (N=100) | Group 3: 30 µg HA + 100 µg LT Patch (N=102) | Group 4: 45 µg HA, no LT Patch (N=50) | Group 5: 45 µg HA + 50 µg LT Patch (N=98) | Group 6: 45 µg HA + 100 µg LT Patch (N=100)
Headache (Nervous system disorders) | 4 | 19 | 13 | 10 | 10 | 9
Malaise (General disorders) | 3 | 13 | 6 | 9 | 9 | 7
Diarrhea (Gastrointestinal disorders) | 4 | 13 | 16 | 4 | 15 | 15
Chills (General disorders) | 0 | 2 | 3 | 3 | 2 | 3
Nausea (Gastrointestinal disorders) | 5 | 11 | 6 | 5 | 12 | 6
Vaccination site erythema (Injury, poisoning and procedural complications) | 2 | 49 | 51 | 3 | 54 | 53
Vaccination site rash (Injury, poisoning and procedural complications) | 0 | 45 | 57 | 2 | 58 | 55
Vaccination site hyperpigmentation (Injury, poisoning and procedural complications) | 0 | 22 | 27 | 0 | 25 | 25
Vaccination site edema (Injury, poisoning and procedural complications) | 1 | 12 | 16 | 1 | 11 | 10
Vaccination site pain (Injury, poisoning and procedural complications) | 7 | 32 | 41 | 13 | 35 | 33
Vaccination site induration (Injury, poisoning and procedural complications) | 6 | 13 | 15 | 8 | 15 | 12
Vaccination site eccymosis (Injury, poisoning and procedural complications) | 1 | 5 | 11 | 1 | 7 | 6
Vaccination site pruritis (Injury, poisoning and procedural complications) | 1 | 45 | 53 | 5 | 51 | 54

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other